CLINICAL TRIAL: NCT04718792
Title: Psilocybin for Treatment of Alcohol Use Disorder: a Feasibility Study
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Anders Fink-Jensen, MD, DMSci (Other)
Collaborators: The Neurobiology Research Unit at Copenhagen University Hospital Rigshospitalet (Unknown)
Responsible Party: Sponsor-Investigator, Anders Fink-Jensen, MD, DMSci, Professor, Psychiatric Centre Rigshospitalet
Organization: Psychiatric Centre Rigshospitalet (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PSILO4ALCO-FEASIBILITY
Record Dates: First submitted 2021-01-08; First posted 2021-01-22 (Actual); Last update posted 2024-07-12 (Actual); Status verified 2024-07

CONDITIONS: Alcohol Use Disorder (AUD)
Keywords: psilocybin; alcohol use disorder; psychedelics; addiction; pharmacokinetics; psilocin; feasibility
MeSH Terms: conditions — Alcoholism; Behavior, Addictive | interventions — Psilocybin

STUDY DESIGN:
Intervention Model Description: Open label study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Psilocybin (Experimental): 10 patients will receive a single administration of psilocybin
  Interventions: Drug: Psilocybin

INTERVENTIONS:
Drug: Psilocybin — A single administration of PEX010 (psilocybin 25 mg, opaque capsule for oral ingestion). PEX010 contains psilocybin (25 mg) naturally extracted from Psilocybe cubensis mushroom fruiting bodies, manufactured under current Good Manufacturing Practices (cGMP)

SUMMARY:
The purpose of this project is to assess the feasibility and safety of administering a single dose of psilocybin to patients diagnosed with alcohol use disorder (AUD). In addition the investigators will establish the pharmacokinetic properties of the active metabolite psilocin. This is the first step in a research project that has the overall aim to evaluate the efficacy of a single administration of psilocybin as an intervention for treatment of AUD.

DETAILED DESCRIPTION:
The investigators will evaluate the feasibility and safety of administering psilocybin to 10 patients diagnosed with AUD. Following informed consent, patients will be screened for eligibility as per in- and exclusion criteria and baseline values will be recorded as per outcome measures. All patients will receive a single administration of 25 mg of psilocybin. As per safety guidelines patients will be monitored the entire dosing session by study staff familiar with the psychedelic effects of psilocybin. In addition, the patients will meet before and after the dosing session with a psychologist connected to the study for preparation and post-session debriefing, respectively. During dosing session, the investigators will collect blood plasma psilocin levels in order to establish pharmacokinetics and an estimated brain 5-HT2AR occupancy. When the effects of psilocybin subside, the investigators will ask the patients to fill out questionnaires encapsulating the psychedelic experience. One week after drug administration the patients are required to meet for an end-of-study assessment of outcome measures including adverse events.

ELIGIBILITY:
Inclusion Criteria:

1. Age of 20-70 years (both included).
2. Body weight of 60-95 kg (both included).
3. Diagnosed with AUD according to DSM-5 criteria and alcohol dependence according to ICD-10.
4. Alcohol Use Disorder Identification Test (AUDIT) ≥ 15.
5. ≥ 5 heavy drinking days.

Exclusion Criteria:

1. Personal or first-degree relatives with current or previous diagnosis within psychotic spectrum disorders or bipolar disorder.
2. History of delirium tremens or alcohol withdrawal seizures.
3. History of suicide attempt or present suicidal ideation.
4. Withdrawal symptoms at inclusion, defined as a score higher than 9 on the Clinical Institute Withdrawal Assessment of Alcohol Scale, Revised (CIWA-Ar).
5. Present or former severe neurological disease including head trauma with loss of consciousness > 30 min.
6. Impaired hepatic function (liver transaminases > 3 times upper normal limit).
7. Cardiac problems defined as decompensated heart failure (NYHA class III or IV), unstable angina pectoris and/or myocardial infarction within the last 12 months.
8. Abnormal electrocardiogram
9. Impaired renal function (eGFR < 50 ml/min).
10. Uncontrolled hypertension (systolic blood pressure >165 mmHg, diastolic blood pressure >95 mmHg).
11. Pharmacotherapy against AUD including disulfiram, naltrexone, acamprosate and nalmefene or treatment with any of these compounds within 28 days prior to inclusion.
12. Treatment with any serotonergic medication or any use of serotonergic psychedelics within 1 month prior to inclusion.
13. Any other active substance use defined as a Drug Use Disorder Identification Test score > 6/2 (m/w) and substance use disorder based on investigator's clinical evaluation, except for nicotine.
14. Women of childbearing potential who are pregnant, breastfeeding or have intention of becoming pregnant or are not using adequate contraceptive measures considered highly effective61.
15. Hypersensitivity to the active substance or to any of the excipients.
16. Unable to speak and/or understand Danish.
17. Any condition that the investigator feels would interfere with trial participation.

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2023-02-09 (Actual); Primary Completion 2024-07-21 (Estimated); Study Completion 2024-07-21 (Estimated)

PRIMARY OUTCOMES:
Safety: Adverse events associated with administration of psilocybin in patients diagnosed with alcohol use disorder | 12 week after drug administration
  Assessment of the incidence and severity of expected and unexpected adverse events

SECONDARY OUTCOMES:
Feasibility: Proportion of participants who complete | 1 week after drug administration
  Proportion of included patients who complete the planned procedures
Pharmacokinetic parameter of psilocin: Cmax | From drug administration and 360 minutes after.
  Cmax: maximum concentration of plasma psilocin determined from concentrations-versus-time data. Blood samples will be drawn with intervals of 20 minutes
Pharmacokinetic parameter of psilocin: Tmax | From drug administration to 360 minutes after.
  Tmax: Time to reach maximum concentration of plasma psilocin determined from concentrations-versus-time data. Blood samples will be drawn with intervals of 20 minutes
Pharmacokinetic parameter of psilocin: AUC | From drug administration to 360 minutes after.
  AUC: Area under the plasma concentrations-versus-time curve determined using the linear trapezoidal rule.
Pharmacokinetic parameter of brain-derived neurotropic factor | From drug administration to 360 minutes after and 1 week after
  Acute and subacute changes in plasma and wholeblod brain-derived neurotropic factor (BDNF)
Pharmacokinetic parameter of cytokines | From drug administration to 360 minutes after and 1 week after
  Acute and subacute changes in plasma cytokines including tumour necrosis factor alpha, interleukin-4 and 6.
Pharmacodynamics of cardiovascular measures | From drug administration to 360 minutes after
  Acute changes in systolic and diastolic blood pressure (mmHg)
Pharmacodynamics of cardiovascular measures | From drug administration to 360 minutes after
  Acute changes in heart rate (beats per minute)
Subjective effects of psilocybin: Intensity | From drug administration to 8 hours after
  Intensity of the drug effect will be assessed with intervals of 20 minutes asking the patients "How intense is the experience right now" on a 0-10 Likert scale where 0 = not intense at all, 10 = very intense.
Subjective effects of psilocybin: Mystical Experience | 8 hours after drug administration
  Experiential aspects of psilocybin measured by The Mystical Experience Questionnaire (MEQ). The patients are asked to rate the items on a 6-point scale going from 0= none; not at all to 5=extreme; more than ever before in my life and stronger than 4.
Subjective effects of psilocybin: Altered States of Consciousness | 8 hours after drug administration
  Experiential aspects of psilocybin measured by the 11-Dimensional Altered State of Consciousness scale (11-DASC). The patients are asked to rate the items by placing marks on a horizontal visual analogue scale (100 millimeters in length) going from "no, not more than usual" (on the left) to "yes, very much more than usual" (on the right).
Subjective effects of psilocybin: Awe Experience | 8 hours after drug administration
  Experiential aspects of psilocybin measured by the Awe Experience Scale. The patients are asked to rate the items on a 7-point scale going from 1= Strongly Disagree to 7= Strongly Agree.
Subjective effects of psilocybin: Ego Dissolution | 8 hours after drug administration
  Experiential aspects of psilocybin measured by the Ego Dissolution Inventory. The patients are asked to rate the items by placing marks on a horizontal visual analogue scale (100 millimeters in length) going from "no, not more than usual" (on the left) to "yes, very much more than usual" (on the right).
Change in heavy drinking days | Baseline, 4, 12 and 52 weeks after drug administration
  Change in heavy drinking day, defined as consuming 60/48 g (men/women) of alcohol or more on any day, in the past 28 days as quantified by the Timeline Followback Method
Change in drinks per day | Baseline, 4, 12 and 52 weeks after drug administration
  Change in drinks per day in the past 28 days as quantified by the Timeline Followback Method
Change in drinking days | Baseline, 4, 12 and 52 weeks after drug administration
  Change in drinking days in the past 28 days as quantified by the Timeline Followback Method
Change in alcohol use | Baseline, 12 and 52 week after drug administration
  Change in self-reported alcohol use measured by the Alcohol Use Identification Test (AUDIT). The AUDIT has 10 questions and the possible responses to each question are scored 0, 1, 2, 3 or 4, with the exception of questions 9 and 10 which have possible responses of 0, 2 and 4. The range of possible scores is from 0 to 40 where 0 indicates an abstainer who has never had any problems from alcoho
Change in craving | Baseline, 1 week, 4 week, 12 and 52 week after drug administration
  Change in self-reported craving measured by the Penn Alcohol Craving Scale (PACS). The patients are asked to rate the items on a 7-point scale going from 0= Never to 6= Nearly all of the time.
Change in self-efficacy | Baseline, 1 week, 4 week, 12 and 52 week after drug administration
  Change in self-reported self-efficacy measured by the Alcohol Abstinence Self-efficacy (AASE). The patients are asked to rate the items on a 5-point scale going from 1= not at all to 5= extremely.
Change in mindfulness | Baseline, 1 week, 4 week, 12 and 52 week after drug administration
  Change in self-reported mindfulness measured by the Mindful Attention Awareness Scale (MAAS). The patients are asked to rate the items on a 6-point scale going from 1= Almost always to 6= Almost never.
Change in psychological flexibility | Baseline, 1 week, 4 week, 12 and 52 week after drug administration
  Change in self-reported flexibility measured by the Acceptance and Action Questionnaire (AAQ). The patients are asked to rate the items on a 7-point scale going from 1= Never true to 7= Always true.
Change in depressive symptoms | Baseline, 1 week, 4 week, 12 and 52 week after drug administration
  Change in self-reported depression symptoms measured by the Major Depressive Inventory (MDI). The patients are asked to rate the items on a 6-point scale going from 1= Always to 7= Never.
Expectancy to treatment | Baseline
  Assessment of the patients expectations before the treatment as measured by the Stanford Expectations of Treatment Scale (SETS).
Persisting Effects | 4, 12 and 52 weeks after drug administration
  Assessment of eight categories of possible changes in attitudes, mood, social effects, and behavior after drug administration
Change in personality traits | Baseline and Week 12 after drug administration
  Change in personality traits as measured by NEO Five-Factor Inventory-3 (NEO-FFI-3). NEO-FFI is 60 items measuring five dimensions of personality: Agreeableness (A), Conscientiousness (C), Neuroticism (N), Extraversion (E), and Openness to Experience (O)

CONTACTS AND LOCATIONS:
Overall Officials: Anders Fink-Jensen, Professor, Principal Investigator — Professor
Locations (1):
- Psychiatric Center Copenhagen, Copenhagen, Frederiksberg, Denmark

REFERENCES:
- [Derived] Jensen ME, Stenbaek DS, Messell CD, Poulsen ED, Varga TV, Fisher PM, Nielsen MKK, Johansen SS, Volkow ND, Knudsen GM, Fink-Jensen A. Single-dose psilocybin therapy for alcohol use disorder: Pharmacokinetics, feasibility, safety and efficacy in an open-label study. J Psychopharmacol. 2025 May;39(5):463-473. doi: 10.1177/02698811251319457. Epub 2025 Feb 28. PMID 40018886